CLINICAL TRIAL: NCT02460211
Title: Acute Effect of Systemic Stress on Measured Blood Concentrations of 25 (OH) Vitamin D
Acronym: ASSESS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1040458
Record Dates: First submitted 2015-04-08; First posted 2015-06-02 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Disease; Vitamin D Deficiency
Keywords: Cardiovascular Disease; Vitamin D; Open Heart Surgery
MeSH Terms: conditions — Cardiovascular Diseases; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Those randomized to the treatment arm will receive three 50,000 unit oral doses of vitamin D3 supplementation.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo/Control Arm (Placebo Comparator): Those randomized to the control arm will receive three oral placebo doses.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Those randomized to the treatment arm will receive three 50,000 unit oral doses of vitamin D3 supplementation. The first dose will be given the evening before surgery. The second and third doses will be given either orally or per NG tube on days 1 and 2 after surgery.
  Arms: Treatment
Dietary Supplement: Placebo — Those randomized to the control arm will receive three placebo doses. The first dose will be given the evening before surgery. The second and third doses will be given either orally or per NG tube on days 1 and 2 after surgery.
  Arms: Placebo/Control Arm

SUMMARY:
Each patient who is admitted for preoperative preparation for elective open heart surgery at Intermountain Medical Center will be invited to participate in this study. After a written informed consent is obtained, patients meeting inclusion/exclusion criteria will be randomized 1:1 to the treatment arm or placebo/control arm. Those randomized to the treatment arm will receive three 50,000 unit oral doses of vitamin D3 supplementation. The first dose will be given the evening before surgery. The second and third doses will be given either orally or per NG tube on the mornings of post-op days 1 and 2. Blood will be obtained at the following time periods: 1) At baseline pre-procedure 12 to 18 hours before planned surgery; 2) Post-operative day 1, 12 to 24 hours after surgery; 3) 48 hours after surgery; 4) 72 hours after surgery; 5) At discharge (estimated to be between 5-8 days after surgery); and 6) At the 6-month follow-up visit (post-surgery). Plasma levels of 25(OH) vitamin D will be measured on each sample.

DETAILED DESCRIPTION:
Each patient who is admitted for preoperative preparation for elective open heart surgery at Intermountain Medical Center will be invited to participate in this study. The patient's history and medical records will be reviewed and data gathered will be used to evaluate the patient's relationship to inclusion and exclusion criteria. After a written informed consent is obtained, subjects will be randomized 1:1 to the treatment arm or placebo/control arm. Those randomized to the treatment arm will receive three 50,000 unit oral doses of vitamin D3 supplementation. The first dose will be given the evening before surgery. The second and third doses will be given either orally or per NG tube on the mornings of post-op days 1 and 2. Approximately 15-20 ml (about one tablespoon) of blood will be obtained at the following time periods (+/- 4 hours): 1) At baseline pre-procedure 12 to 18 hours before planned surgery; 2) Post-operative day 1, 12 to 24 hours after surgery; 3) 48 hours after surgery; 4) 72 hours after surgery; 5) At discharge (estimated to be between 5-8 days after surgery); and 6) At the 6-month follow-up visit (post-surgery). Each blood sample will be transported to The Center for Molecular and Genetic Research at LDS Hospital Cardiovascular Genetics Laboratory for preparation and storage. Plasma levels of 25(OH) vitamin D will be measured on each sample.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >= 18 years of age
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures
3. Subject is scheduled for elective open heart surgery at Intermountain Medical Center
4. Subject is relatively stable as assessed by the Principal Investigator

Exclusion Criteria:

1. Inability or refusal of the patient and/or the patient's legally acceptable representative to provide written informed consent for any reason.
2. History of previous vitamin D supplementation > 1,000 units of vitamin D3 per day within the past three months.
3. Evidence of hypercalcemia on screening labs (> 10.5 milligrams per deciliter of blood).
4. Any scheduled cardiac surgical procedure that does not require open thoracotomy (the reason for this exclusion is that the study design requires that the patients will undergo a significantly stressful procedure, which can be generally guaranteed if the patient undergoes open thoracotomy).
5. Known allergic reaction or other intolerance to oral vitamin D3.
6. Pregnant and/or lactating women and women of child bearing potential who are not using acceptable means of contraception. Women of childbearing potential must be using adequate measures of contraception (as determined by the Principal Investigator) to avoid pregnancy and should be highly unlikely to conceive during the study period. Women of childbearing potential must have a negative pregnancy test at screen.
7. Subject participation in previous investigational interventional studies within 30 days of the current study.
8. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in 25(OH) vitamin D levels (ng/ml) between baseline (pre-surgery) and 72 hours post-surgery. | 72 hours

SECONDARY OUTCOMES:
Comparison of 25(OH) vitamin D levels (ng/ml) between baseline and other time points. | 12-24 hrs, 48 hrs, discharge (approximately 5-8 days post-surgery), 6 months
  Subjects will be re-assessed on post-operative day 1 (12-24 hours after surgery), then at 48 and 72 hours post-surgery, at discharge (approximately 5-8 days post-surgery), and at a 6 month post-surgery follow-up visit.
Percent differences in adverse clinical outcomes between the vitamin D3 supplementation treatment and placebo arms. | 6 months
  Clinical outcomes that will be monitored include: death, myocardial infarction, stroke, repeat coronary revascularization or hospitalization for heart failure, worsening of renal function, hospitalization for pneumonia or other acute systemic infection or any other serious adverse clinical event.
Time to adverse clinical events stratified by vitamin D3 supplementation and placebo arms. | 6 months
  Clinical outcomes that will be monitored include: death, myocardial infarction, stroke, repeat coronary revascularization or hospitalization for heart failure, worsening of renal function, hospitalization for pneumonia or other acute systemic infection or any other serious adverse clinical event.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Muhlestein, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States

REFERENCES:
- [Derived] Barker T, May HT, Doty JR, Lappe DL, Knowlton KU, Carlquist J, Konery K, Inglet S, Chisum B, Galenko O, Anderson JL, Muhlestein JB. Vitamin D supplementation protects against reductions in plasma 25-hydroxyvitamin D induced by open-heart surgery: Assess-d trial. Physiol Rep. 2021 Feb;9(3):e14747. doi: 10.14814/phy2.14747. PMID 33580636